CLINICAL TRIAL: NCT05097001
Title: Dystonia Image-based Programming of Stimulation: A Prospective, Randomized, Double-blind Crossover Trial
Acronym: DIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: BMBF (Bundes Ministerium fuer Bildung und Forschung) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DIPS
Record Dates: First submitted 2021-10-01; First posted 2021-10-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Dystonia; Deep Brain Stimulation
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer (Experimental): Programming based on computer-guided assessment
  Interventions: Other: DBS programming
- CLINICAL (Active Comparator): Programming based on clinically-guided assessment
  Interventions: Other: DBS programming

INTERVENTIONS:
Other: DBS programming — DBS readjustment based on COMPUTER or CLINICAL program

SUMMARY:
The primary objective of this exploratory study is to prospectively evaluate the feasibility of image-guided programming of pallidal deep brain stimulation (DBS) for dystonia. The dystonias are a heterogeneous group of movement disorders that share the core clinical feature of abnormal involuntary muscle contractions in common. Pallidal DBS is an established therapy for severe cases with an average improvement in dystonia severity of 50-60%. However, outcomes are variable and difficult to predict, and clinical trials report up to 25% of Nonresponders. Variability in electrode placement and inappropriate stimulation settings may account for much of this variability in outcome. In addition, improvement in dystonia is delayed, often days to weeks after a change in DBS therapy, complicating programming.

Our group recently developed a computer model to predict optimal individualized stimulation settings in patients based on the outcome of a large cohort of of chronically treated patients. In-silico testing showed a 16.3% better mean group improvement with computer-assisted programming compared with physician-assisted programming and a dramatic reduction in non-responders (from 25% to 5%).

In this prospective study, the computer model will be compared in a randomized, controlled, and double blinded setting against best clinical DBS programming. The primary outcome will be a responder analysis in which dystonia severity will be compared between conventional clinical and model-based programming will be compared.

DETAILED DESCRIPTION:
Dystonia is a neurological syndrome characterized by involuntary, sustained, or repetitive muscle contractions of opposing muscle groups that cause twisting movements and abnormal postures. Dystonias meet the prevalence criterion of a rare disorder, with prevalence estimates ranging from 0.2-5/100,000 for infantile or juvenile forms to 3-732/100,000 for dystonias manifesting in adults. In addition to motor impairments and mobility limitations, patients - especially young patients - suffer from non-motor symptoms: depression (> 15%), anxiety (> 25%), decreased sleep quality (> 70%), and pain (> 75%). In addition, there is a high risk of economic impairment, including job loss (> 55%), and decreased productivity are serious social consequences (> 50%). However, disability is usually secondary to motor impairment, and adequate treatment of motor symptoms can lead to profound improvements in quality of life (Skogseid et al. 2007). Currently, there is no cure for dystonia, and pharmacological symptom treatment is limited. Deep brain stimulation (DBS) of the internal globus pallidus (GPi) is a recommended therapy for severe dystonia with Class I evidence for safety and efficacy (Vidailhet et al. 2005; Volkmann et al. 2012; Volkmann et al. 2014). However, clinical trials report up to 25% non-responders (<25% motor improvement) (Volkmann et al. 2012; Volkmann et al. 2014). Variability in electrode placement and inappropriate stimulation settings may explain much of this outcome variability (Reich et al. 2019). In addition, dystonia improves with a delay, often weeks after initiation or days after switching neurostimulation therapy, complicating clinical programming for DBS (Kupsch et al. 2011). Our group recently presented a novel approach based on empirical knowledge from a large cohort of chronically treated patients. We defined probabilistic maps of antidystonic effects using electrode position and volumes of tissue activation (VTA) from >100 patients. This method predicts a 16.3% better mean group improvement with computer-selected electrode choices compared with physician programming and a reduced proportion of non-responders from 25% to <5% (Reich et al. 2019). This potential advantage of computer-assisted programming capabilities will be tested in the study described here.

This study is supported by the Bundesministerium für Bildung und Forschung (BMBF): Förderkennzeichen: 01KG2032

ELIGIBILITY:
Inclusion Criteria:

* Chronic deep brain stimulation (> 1 year) in the internal globus pallidus in patients with isolated dystonia.
* Deep brain stimulation settings and dystonia medication stable for > 3 months.
* Understanding about and consent to the study and signed informed consent form.

Exclusion Criteria:

* Relevant comorbidities that might interfere with study endpoints (esp. palliative disease and severe neurologic or psychiatric comorbidities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
successful treatment with model predicted settings | 8 week follow-up
  The primary efficacy endpoint is based on the blinded physician rating of dystonia severity reflected by Clinical Dystonia Rating Scales (BFMDRS or TWSTRS). The raters will be internationally recognized leading experts in the field of movement disorders that are not part of the study team or otherwise related to our center. For both interventions (best clinical settings and model predicted settings) we will calculate the symptom severity score after 4 weeks of continuous stimulation, expressed in percent of the pre-operative score. The primary endpoint is defined as "successful treatment with model predicted settings" (yes or no). The value is "yes" if the motor symptoms with model predicted settings are equal or better (tolerance 5%) to clinical settings.

SECONDARY OUTCOMES:
quality of life SF-36 (Short Form-36) | 4 week and 8 week follow-up
  SF-36 questionnaire (Short Form-36): 36 items [0-36 points, the higher the score, the worse the symptoms]
quality of life CDQ24 | 4 week and 8 week follow-up
  CDQ24 questionnaire (Craniocervical dystonia questionnaire 24): 24 items [0-24 points, the higher the score, the worse the symptoms]
calculated energy consumption | Baseline visit
  Energy consumption by the DBS pulse generators
time for programming | Baseline visit
  Time necessary to program the optimal DBS settings

CONTACTS AND LOCATIONS:
Overall Officials: Martin Reich, Principal Investigator — Department of Neurology - University Hosiptal Würzburg
Locations (1):
- Department of Neurology, University Hospital Würzburg, Würzburg, Bavaria, Germany

REFERENCES:
- [Derived] Lange F, Roothans J, Wichmann T, Gelbrich G, Roser C, Volkmann J, Reich M. DIPS (Dystonia Image-based Programming of Stimulation: a prospective, randomized, double-blind crossover trial). Neurol Res Pract. 2021 Dec 20;3(1):65. doi: 10.1186/s42466-021-00165-6. PMID 34924027